CLINICAL TRIAL: NCT02878993
Title: Predicting Infant Extubation Using Diaphragm Surface Electromyography
Acronym: EMG
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: KCH16-100; 16/LO/1281 (Other: NHS REC); 205807 (Other: IRAS)
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2018-03

CONDITIONS: Infant, Newborn, Disease
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intubated infants: Recording of diaphragm EMG
  Interventions: Device: Recording of diaphragm EMG

INTERVENTIONS:
Device: Recording of diaphragm EMG — Recording of diaphragm EMG prior to extubation using surface diaphragm electromyography

SUMMARY:
This study aims to assess whether the electrical signal of the diaphragm (diaphragm electromyogram) and the ratio of that to tidal volume (amount of air breathed in and out of the lungs) can predict which infants will be successfully extubated (have the breathing tube removed without needing it replaced.)

DETAILED DESCRIPTION:
This study aims to assess whether the electrical signal of the diaphragm (diaphragm electromyogram) and the ratio of that to tidal volume (amount of air breathed in and out of the lungs) can predict which infants will be successfully extubated (have the breathing tube removed without needing it replaced.)

ELIGIBILITY:
Inclusion Criteria:

* intubated and mechanically ventilated on NICU

Exclusion Criteria:

* major congenital abnormalities

Ages: 0 Days to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants mechanically ventilated on NICU without major congenital abnormalities
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2016-08; Primary Completion 2018-05 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Magnitude of diaphragm EMG | One hour
  Magnitude of diaphragm EMG
Ratio of diaphragm EMG to tidal volume | One hour
  Ratio of diaphragm EMG to tidal volume

SECONDARY OUTCOMES:
Extubation success | 48 hours
  Extubation success is define as remaining free of invasive mechanical ventilation. Whether the above measures of diaphragm EMG can predict such success will be investigated

CONTACTS AND LOCATIONS:
Overall Officials: Anne Greenough, Principal Investigator — King's College London
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hunt KA, Hunt I, Ali K, Dassios T, Greenough A. Prediction of extubation success using the diaphragmatic electromyograph results in ventilated neonates. J Perinat Med. 2020 Jul 28;48(6):609-614. doi: 10.1515/jpm-2020-0129. PMID 32598319